CLINICAL TRIAL: NCT04887467
Title: Pharmacokinetic Study of Continuous and Diurnal Subcutaneous Apomorphine Infusion in Patients With Parkinson's Disease Under Stabilized Treatment.
Brief Title: Monocentric, Prospective Study to Assess the Pharmacokinetic Profile of Continuous and Diurnal Subcutaneous Apomorphine Infusion in Patients With Parkinson's Disease
Acronym: PHARM-APO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35RC21_9909_PHARM-APO
Record Dates: First submitted 2021-04-26; First posted 2021-05-14 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
Keywords: Apomorphine; Pharmacokinetics; Dopamine Agonists
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Parkinson disease (Experimental): Apomorphine 5mg/mL, solution for infusion, intraveinous use
  Interventions: Drug: Apomorphine

INTERVENTIONS:
Drug: Apomorphine — Assigned Interventions:
  * blood sampling
  * blood collection
  * systolic, diastolic, mean blood pressure and heart rate measure

SUMMARY:
This monocentric and prospective trial aims firstly to assess the pharmacokinetic profile of continuous and diurnal subcutaneous apomorphine infusion in patients with Parkinson's disease under stabilized treatment and, secondly, to collect data highlighting the possible influence of pharmacogenetics.

DETAILED DESCRIPTION:
A screening visit will be conducted 15 days to 2 months prior to the patient's hospitalization. Each subject will undergo a clinical examination including a collection of data relating to medical and surgical history, specific data related to Parkinson's disease and apomorphine pump treatment, and the completion of all items of the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) 3 scale in ON condition. Verification of the biological parameters necessary for the proper conduct of a pharmacokinetic study will also be carried out (venous capital; search for possible hepatic and/or renal failure).

The subjects will be called to the hospital two by two at 4:00 pm for a medical visit, during which a clinical examination will be performed (height, weight, fat mass, occurrence of infectious and/or inflammatory episodes) The subjects will then be placed in a room. A catheter will be placed in a forearm vein to allow blood sampling. All plasma samples will be taken from subjects who have been supine for at least 30 minutes. Blood pressure and heart rate will be checked before each sample.

A first blood sample will be taken at 8 pm followed by a standardized dinner. After the pump is stopped and removed at the patient's usual time, consecutive blood samples will be taken at T30, T60, T120, and T180 (i.e., 30 min, 1 h, 2 h, and 3 h after pump removal). The next morning, a new blood sample will be taken 10 min before the pump is turned on, at the usual time. A standardized breakfast will be served. A new series of consecutive blood samples will be taken at T30, T60, T120 and T180, following the same pattern as before.

A standardized lunch will be served around 11:30 am, and the patients will be allowed to leave after medical advice, at the latest at 2 pm.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 70 year-old males
* Suffering from Parkinson's disease, considered to be well controlled by treatment, including apomorphine (CGI criteria)
* Use of daytime apomorphine pump treatment (nighttime discontinuation) for a minimum of 6 months, with a good tolerance and treatment dosage unchanged for a minimum of 3 months (apomorphine flow rate and daily dose and oral concomitant antiparkinsonian medication if applicable)
* Autonomous patient in the apomorphine pump daily management (start and removal)
* Written informed consent
* Restrictive criteria to limit confounding factors : apomorphine type (Apokinon® apomorphine, cartridge or ampoule, Aguettant pharmaceutical laboratory) and medical device (Microjet CRONO-PAR pump (N=10) and France Développement Electronique (FDE) So Connect pump (N=10))

Exclusion Criteria:

* Concomitant participation in a clinical trial that may affect the biological and/or pharmacokinetic parameters
* Clinically relevant hepatic dysfunction that may significantly alter drug metabolism (value >2 times the upper limit of normal)
* Clinically relevant renal dysfunction that may significantly alter drug excretion (clearance < 30 mL/min (chronic renal failure))
* Alcohol abuse (> 30 g pure alcohol per day*) or drug addiction
* Current tobacco consumption ; for ex-smokers : stopping smoking for less than 1 month at the time of inclusion
* Dementia or cognitive impairment considered clinically significant
* Adults legally protected (under judicial protection, guardianship or supervision), persons deprived of their liberty

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Area under the curve of plasma apomorphine concentration between 0h and 24h | up to 24 hours

SECONDARY OUTCOMES:
Systolic blood pressure variations measured prior to each blood collection | up to 24 hours
Diastolic blood pressure variations measured prior to each blood collection | up to 24 hours
Mean blood pressure variations measured prior to each blood collection | up to 24 hours
Heart rate variations measured prior to each blood collection | up to 24 hours
Area under the curve of plasma apomorphine concentration - time values curve from treatment administration (t0) until 6h after (AUC0-6) | up to 24 hours
Half-life (t1/2) determined by the t1/2 = Ln2/λz formula | up to 24 hours
Apparent total clearance (Cl/F) and apparent volume of distribution (Vd) calculated according to the formulas Cl/F = Dose/AUC0-24 et Vd = Cl(T)/λz wherein F is the absolute bioavailability | up to 24 hours
Study of weight on area under the curve of drug concentrations | up to 24 hours
Study of liver function on area under the curve of drug concentrations | up to 24 hours
Study of the main genes involved in the biotransformation and transport of apomorphine | up to 24 hours
  DNA bank
Study of the pump type on area under the curve of drug concentrations | up to 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Pontchaillou, Rennes, France

IPD SHARING:
Plan to Share IPD: No